| Participant No: | Date: |
|-----------------|-------|
|-----------------|-------|



## Department of Psychiatry | The University of Hong Kong

## **Informed Consent Form**

## The effectiveness of rTMS on improving food cravings and weight control in adults without serious mental illness

Principal Investigator: Dr. Cheng Pak Wing, Assistant Professor, Department of Psychiatry, Faculty of Medicine, The University of Hong Kong

| 1 | The participant has read and understood the information sheet for the study dated//, and have had the opportunity to ask questions. | | |
|---|---|---|---|
| 2 | The participant understands that participation is voluntary, and that one may withdraw at a time without providing any reason, and without affecting our medical care or legal rights. | | |
| 3 | The participant understands that in relation to this study, personnel from the Department of Psychiatry of The University of Hong Kong, The University of Hong Kong itself, the Institutional Review Board of the University of Hong Kong/ Hospital Authority Hong Kong West Cluster, or regulatory authorities may access the participant's medical records. The participant gives permission for such individuals to access these records. | | |
| 4 | The participant is required to undergo six sessions of repetitive transcranial magnetic stimulation (rTMS) and gives permission/authorization for researchers to administer the rTMS. | | |
| 5 | The participant agrees that the researchers may contact us in the future using the contact details provided in this study for related research purposes. | | |
| 6 | 6 All procedures involved in the study are provided free of charge. | | |
| 7 | There are no conflicts of interest regarding the use of the rTMS machine in this study that influenced the design, implementation, or interpretation of the research. | | |
| Nam | e of Participant | Date | Signature |
| Name of Researcher | | Date | Signature |